CLINICAL TRIAL: NCT05953935
Title: Effect Of Resistive Capactive Electrical Transfer Therapy On Wound Healing And Biomarker Expression In Difficult-to-heal Wounds
Brief Title: Effect Of Resistive Capactive Electrical Transfer Therapy In Difficult-to-heal Wounds
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CRET-ÚLCERAS-01
Record Dates: First submitted 2023-06-29; First posted 2023-07-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Difficult-to-heal Wounds

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, randomized, interventional, pre-post clinical study with control group and seamless adaptive design. It will be conducted in two phases: 1) exploratory phase (E) and 2) confirmatory phase (C), depending on the results obtained in the exploratory phase. Patients will be randomized to control group (standard clinical procedures) and experimental group (OKTO medical device)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A-E group (Experimental): Treatment with radiofrequency currents of resistive capacitive electrical transfer therapy (CRET) under hyperthermia conditions plus standard clinical treatments, in patients with ulcers of venous etiology.
  Interventions: Device: OKTO; Device: Standard clinical procedures
- B-E group (Experimental): Treatment with radiofrequency currents of resistive capacitive electrical transfer therapy (CRET) under hyperthermia conditions plus standard clinical treatments in patients with diabetic foot ulcers.
  Interventions: Device: OKTO; Device: Standard clinical procedures
- A-C grouop (Experimental): Treatment with radiofrequency currents of resistive capacitive electrical transfer therapy (CRET) under hyperthermia conditions plus standard clinical treatments in CDH.
  Interventions: Device: OKTO; Device: Standard clinical procedures
- B-C grouop (Experimental): Treatment with radiofrequency currents of resistive capacitive electrical transfer therapy (CRET) under subthermal conditions plus standard clinical treatments in CDH.
  Interventions: Device: OKTO; Device: Standard clinical procedures
- C-C group (Experimental): Standard clinical treatments established on the basis of the treatment standards of the International Working Group on the Diabetic Foot (IWGDF), in the case of diabetic foot ulcers (2, 3). For ulcers of venous etiology, the treatment standards according to the guidelines of the Spanish Association of Vascular Nursing and Wounds (Asociación Española de Enfermería Vascular y Heridas) will also be applied.
  Interventions: Device: Standard clinical procedures

INTERVENTIONS:
Device: OKTO — Static Monopolar Capacitive Resistive Resistive Radiofrequency Equipment at 448 kHz
  Arms: A-C grouop; A-E group; B-C grouop; B-E group
Device: Standard clinical procedures — standard clinical procedures

SUMMARY:
Difficult-to-heal wounds present imbalances in cytokine production, increases in MMP expression, high levels of apoptosis, and decreases in the proliferation of cells such as fibroblasts and keratinocytes, which are involved in tissue regeneration. CRET therapy (capacitive resistive electrical transfer therapy) has been shown to generate granulation tissue in in vitro assays. In addition, available clinical case reports and preliminary clinical trial results indicate that CRET can promote the regeneration of acute wounds and DHW (difficult-to-heal wounds).

DETAILED DESCRIPTION:
Difficult-to-heal wounds present imbalances in cytokine production, increases in MMP expression, high levels of apoptosis, and decreases in the proliferation of cells such as fibroblasts and keratinocytes, which are involved in tissue regeneration. CRET therapy has been shown to be able to generate granulation tissue in in vitro assays. In addition, available clinical case reports and preliminary clinical trial results indicate that CRET can promote acute wound regeneration and CDH.

The working hypothesis is that CRET treatment promotes the healing of CDH through its action in regulating inflammatory and regenerative processes in skin tissue. This non-invasive, cost-effective treatment, devoid of identified adverse effects, and not studied in depth so far in patients with CDH, can thus be placed in the treatment algorithms of CDH with the correct selection of candidate patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Agree to participate in the study and sign the informed consent form.
* Inpatients or outpatients who can be followed by the research team for the duration of the study
* Ulcers with a surface area of no less than 0.5 cm2 and of at least 4 weeks' duration (CDH), located on the lower limbs in the case of ulcers of venous etiology or on the foot, in the case of diabetic foot ulcers.
* For patients with ulcers of venous etiology: ulcers of venous etiology stage 2, 3 4 with diagnosis of chronic venous insufficiency with open wound CEAP IVC C6 according to CEAP classification (38).
* For patients with diabetic foot ulcers presenting:

  * Type 1 and type 2 diabetics with a glycated hemoglobin (HbA1c ≤10% (in a test no longer than 3 months).
  * Patients with UPD without PAD or with associated mild or moderate stage PAD (39) according to the criteria of the intersociety consensus for the treatment of peripheral arterial disease (TASC II).
  * UPD Grade 1A, 1C, 2A, 2C according to the Texas classification (40).
  * Patients who have required previous surgical debridement and 4 weeks have elapsed since such debridement.
* Comorbidity is defined as the presence of at least one of the following criteria:

  * Smoking more than 10 cigarettes per day in the last 6 months.
  * Immunosuppression: systemic treatment with high-dose corticosteroids in the previous 3 months, severe active infection in the previous month, presence of systemic or organ-specific autoimmune disease.
  * Renal failure with creatinine > 2 mg/dl.
  * Respiratory failure with pO2< 90 mm Hg
  * Cardiac failure, grade II or higher
  * Anemia or nutritional deficit
  * Endocrine disruption under medical treatment
  * Neuropathy in the affected area or neurological disease.
  * Connective tissue diseases
  * Mobility impairment
  * Presence of microvascular disease

Exclusion Criteria:

* Pregnancy
* Patients with contraindications for CRET treatments (electronic implants, thrombophlebitis).
* Patients with chronic or pathological wounds that required surgical intervention.
* Ulcers with active infection according to IDSA classification in soft tissues or with clinical and/or radiological signs compatible with osteomyelitis.
* Allergies to standard wound treatment.
* Patients presenting severe renal insufficiency (Glomerular filtration rate ≤30 ml/min in analysis performed in the last 3 months).
* Patient who has presented an acute ischemic event (acute myocardial infarction or stroke, in the 3 months prior to inclusion in the study).
* Patients who present an evolving neoplastic condition, treated by radiotherapy, chemotherapy, hormone therapy or immunosuppressants at the current moment.
* Patients treated for a chronic condition requiring the intake of strong systemic corticosteroids doses ≥ 40 mg prednisone).
* Critical non-revascularizable ischemia or TcPO2 < 25mmHg or a digital hallux systolic pressure < 50 mm Hg in diabetic foot ulcers.
* Patients who do not accept to use the prescribed unloading treatment in the case of diabetic foot ulcers.
* In the case of patients with ulcers of venous etiology, the presence of peripheral arterial disease in any of its stages.
* Patients who do not accept the indicated compressive bandage treatment, in the case of ulcers of venous etiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Wound dimensions before and after treatments in patients with HDC treated with CRET therapy plus standard treatment versus patients with HDC undergoing standard treatment alone. | 18 months
  Wound dimensions measurement (area, length and width) before and after treatments in patients with HDC treated with CRET therapy plus standard treatment versus patients with HDC undergoing standard treatment alone.

SECONDARY OUTCOMES:
General clinical evaluation: | 18 months
  * age,
  * sex,
  * BMI
  * general medical history,
  * baseline blood work,
  * usual treatment
Wound evaluation: | 18 months
  * cause,
  * location,
  * time of evolution,
  * photographs.
Evaluation of biomarkers in peripheral blood of patients with CDH with or without CRET treatment: | 18 months
  Quantification of cytokines and growth factors: IL-1α, IL-1β, TNFα, IFγ.
In primary cultures of fibroblasts isolated from biopsies of CDH patients with or without CRET treatment, assessment of typical CDH biomarkers related to: | 18 months
  * Death: TUNEL assay; Bcl-2, Bcl-X and Caspase-3 markers.
  * Viability/proliferation: XTT, Ki67, p-p38 and p-ERK1/2 assays.
  * Adhesion: β -catenin and E-cadherin.
  * Extracellular matrix: α-SMA, Col I and Col III and the metalloproteinases, MMP8, MMP2 and MMP9.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Hernández Bule, PhD, Principal Investigator — IRYCIS. Hospital Universitario Ramón y Cajal. Madrid, Spain.
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No